CLINICAL TRIAL: NCT00553735
Title: The Prophylactic Use of Topical Cyclosporine A 0.05% (Restasis) to Prevent Onset and Progression of Graft-versus-host Disease-related Dry Eye
Brief Title: The Prophylactic Use of Topical Cyclosporine A 0.05% to Prevent Graft Versus Host Disease Related Dry Eye
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: High number of withdrawals, appt. no-shows, or those lost to follow-up.
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: 07-05-034; 07-05-034 (Other: Massachusetts Eye and Ear)
Record Dates: First submitted 2007-11-02; First posted 2007-11-06 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2013-04

CONDITIONS: Dry Eye
Keywords: Dry Eye; Graft versus Host Disease; GVHD
MeSH Terms: conditions — Dry Eye Syndromes; Graft vs Host Disease | interventions — Cyclosporins; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cyclosporine A 0.05% (Active Comparator): If patients pass the screening criteria, both eyes are randomized to therapy. One eye will receive Cyclosporine A 0.05% (Restasis) and the other eye will receive Placebo (Artificial Tear)
  The objective signs will be corneal and conjunctival staining, Schirmer test (with and without anesthesia), and tear break-up time. The subjective endpoints will be the SANDE symptom global score.
  Interventions: Drug: Cyclosporine A 0.05%
- Artificial Tear (Placebo Comparator): If patients pass the screening criteria, both eyes are randomized to therapy. One eye will receive Cyclosporine A 0.05% (Restasis) and the other eye will receive Placebo (Artificial Tear)
  The objective signs will be corneal and conjunctival staining, Schirmer test (with and without anesthesia), and tear break-up time. The subjective endpoints will be the SANDE symptom global score.
  Interventions: Drug: Arificial Tear

INTERVENTIONS:
Drug: Cyclosporine A 0.05% — Topical cyclosporine A 0.05% (Restasis) three times a day for 18 months.
  Other Names: Restasis
  Arms: Cyclosporine A 0.05%
Drug: Arificial Tear — Artificial Tear - three times a day for 18 months.
  Other Names: Placebo; Artificial Tear
  Arms: Artificial Tear

SUMMARY:
The purpose of this study is to determine whether Restasis is an effective treatment for preventing the occurrence and progression of dry eye syndrome in patients who have recently received a bone marrow transplant and are at risk to graft-versus-host disease.

DETAILED DESCRIPTION:
The purpose of this research study is to determine if early treatment using Restasis eye drops can prevent the development or delay the progression of dry eye syndrome in allogeneic bone marrow transplant (BMT) recipients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* At least 18 years of age
* Approved candidate for allogeneic HSCT
* Ability to understand and provide informed consent to participate in this study
* Willingness to follow study instructions and likely to complete all required visits

Exclusion Criteria:

* History of ocular or eyelid surgery
* History of glaucoma or ocular hypertension
* History of herpetic eye disease
* Patient with acne rosacea, blepharitis, or meibomitis, in the opinion of the investigator
* Any ocular disorder or condition (including ocular infection, trauma, and disease) that could possibly interfere with the interpretation of the study results
* Recent (3-month) history of wearing contact lens
* Anticipated contact lens wear during any portion of the study
* Recent (3-month) history of current use of topical steroids or antiglaucoma agents
* Any punctal occlusion within 2 months of the screening visit
* Significant sign or symptoms of dry eye (the definition of "dry eye" used for exclusion criteria is compatible with the recommendations of the NEI/Industry Workshop on Clinical Trials in Dry Eyes (Lemp, 1995) (see Appendix 1and 2))
* History of connective tissue disease or diabetes
* Any condition (including language barrier) that precludes patient's ability to comply with study requirements including completion of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reza Dana, M.D., Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: Each eye of every participant was randomized to therapy. One eye will receive Cyclosporine A 0.05% (Restasis) and the other eye will receive placebo (Artificial Tear)
  The objective signs will be corneal and conjunctival staining, Schirmer test (with and without anesthesia), and tear break-up time. The subjective endpoints will be the SANDE symptom global score.
  Cyclosporine A 0.05% : Topical cyclosporine A 0.05% (Restasis) three times a day for 18 months.
Period: Overall Study
Arm/Group | All Study Participants
Started | 8
Completed | 1
Not Completed | 7

BASELINE CHARACTERISTICS:
Groups:
- Arm I: The objective signs will be corneal and conjunctival staining, Schirmer test (with and without anesthesia), and tear break-up time. The subjective endpoints will be the SANDE symptom global score.
  Cyclosporine A 0.05% : Topical cyclosporine A 0.05% (Restasis) three times a day for 18 months.
Arm/Group | Arm I
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Corneal Staining Score
Time Frame: 18 months
Population: No data were collected because participants withdrew themselves, failed to show for their appointments, or were lost to follow-up.
Groups:
- Cyclosporine A 0.05%: If patients pass the screening criteria, both eyes are randomized to therapy. One eye will receive Cyclosporine A 0.05% (Restasis) and the other eye will receive Placebo (Artificial Tear)
  The objective signs will be corneal and conjunctival staining, Schirmer test (with and without anesthesia), and tear break-up time. The subjective endpoints will be the SANDE symptom global score.
  Cyclosporine A 0.05%: Topical cyclosporine A 0.05% (Restasis) three times a day for 18 months.
- Artificial Tear: If patients pass the screening criteria, both eyes are randomized to therapy. One eye will receive Cyclosporine A 0.05% (Restasis) and the other eye will receive Placebo (Artificial Tear)
  The objective signs will be corneal and conjunctival staining, Schirmer test (with and without anesthesia), and tear break-up time. The subjective endpoints will be the SANDE symptom global score.
  Arificial Tear: Artificial Tear - three times a day for 18 months.
Arm/Group | Cyclosporine A 0.05% | Artificial Tear
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Conjunctival Staining Score
Time Frame: 18 Months
Population: as for outcome 1
Arm/Group | Cyclosporine A 0.05% | Artificial Tear
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Incidence and Severity of Ocular Adverse Event
Description: Incidence and severity of ocular adverse events, as identified by eye examination and visual acuity testing.
Time Frame: 18 Months
Population: All patients enrolled in the study were analyzed.
Measure: Number; unit: participants
Groups:
- Cyclosporine A 0.05%: The objective signs will be corneal and conjunctival staining, Schirmer test (with and without anesthesia), and tear break-up time. The subjective endpoints will be the SANDE symptom global score.
  Cyclosporine A 0.05% : Topical cyclosporine A 0.05% (Restasis) three times a day for 18 months.
- Artificial Tear: The objective signs will be corneal and conjunctival staining, Schirmer test (with and without anesthesia), and tear break-up time. The subjective endpoints will be the SANDE symptom global score.
  Artificial Tear three times a day for 18 months.
Arm/Group | Cyclosporine A 0.05% | Artificial Tear
Number analyzed (Participants) | 8 | 8
participants | 2 | 2

4. Secondary Outcome: Symptom Assessment iN Dry Eye (SANDE) Patient Questionnaire
Time Frame: 18 Months
Population: as for outcome 1
Arm/Group | Cyclosporine A 0.05% | Artificial Tear
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Tear Break-up Time (TBUT)
Time Frame: 18 Months
Population: as for outcome 1
Arm/Group | Cyclosporine A 0.05% | Artificial Tear
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Schirmer Without Anesthesia
Time Frame: 18 Months
Population: as for outcome 1
Arm/Group | Cyclosporine A 0.05% | Artificial Tear
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Schirmer With Anesthesia
Time Frame: 18 Months
Population: as for outcome 1
Arm/Group | Cyclosporine A 0.05% | Artificial Tear
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The adverse events reported are by "eye". Two adverse events were reported: uveitis and bacterial infection. Both these events were bilateral (i.e. both eyes), occurring in two separate subjects.
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=8)
Uveitis (bilateral) (Eye disorders) | 1 (1)
Bacterial Infection (bilateral) (Eye disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated early due to a high number of patients who withdrew themselves, failed to show for their appointments, or were lost to follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No